CLINICAL TRIAL: NCT01197859
Title: Three Month Clinical Evaluation of the Contamac 74% Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contamac Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCSH-1901
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Vision Correction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Contamac 74% silicone hydrogel contact lens (Active Comparator): Definitive Contact Lens
  Interventions: Device: Definitive Contact Lens
- Cooper Vision Biofinity (Placebo Comparator): Biofinity Contact Lens
  Interventions: Device: Biofinity

INTERVENTIONS:
Device: Definitive Contact Lens — Daily wear contact lens
  Arms: Contamac 74% silicone hydrogel contact lens
Device: Biofinity — Daily wear contact lens
  Arms: Cooper Vision Biofinity

SUMMARY:
The purpose of this study is to compare the clinical performance of the contamac silicone hydrogel contact lens with a predicate device (Cooper Vision Biofinity).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the clinical performance of the Contamac lens in comparison with a currently marketed silicone hydrogel: Biofinity® (CooperVision). This is a 3-month, open-label, bilateral, parallel group, randomised, daily wear study. Approx. two-thirds of the subjects will wear the Contamac Silicone Hydrogel lens in both eyes while the other third will wear control lenses.

ELIGIBILITY:
Inclusion Criteria:

* existing contact lens wearer
* read and signed statement of informed consent
* has clear central cornea
* requires spherical distance correction

Exclusion Criteria:

* has worn RGP contact lenses within the last 30 days
* is using any ocular medication
* has had refractive surgery
* has an infectious disease
* is pregnant or lactating
* is participating in another clinical research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Assess performance variables as compared to the predicate device during follow-up visits to demonstrate safety and efficacy. | 3 months
  The clinical study will assess the following performance variables as compared to the predicate device during 5 follow-up visits over a 3 month period to demonstrate safety and efficacy: Sphere-cyl Refraction and VA, Keratometry, Comfort, Handling, Symptoms, Over-Refraction and VA, Lens Fit, Lens Deposits, and Slit Lamp Findings.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, Principal Investigator — Vision Care Research
Locations (1):
- Vision Care Research, Farnham, Surry, United Kingdom